CLINICAL TRIAL: NCT07368166
Title: Development of the PTSD-iMPACT to Measure PTSD-Related Functional Impairment in Children and Adolescents - A Validation Study in Switzerland and Germany
Acronym: PTSD-iMPACT
Status: Recruiting | Type: Observational
Sponsor: University Children's Hospital, Zurich (Other)
Collaborators: University Clinic for Child and Adolescent Psychiatry, Psychosomatics, and Psychotherapy, Carl von Ossietzky University of Oldenburg, Oldenburg, Germany (Unknown); Outpatient clinic for trauma, Clinic for Psychiatry, Psychosomatics, and Psychotherapy for Children and Adolescents, RHTW Aachen, Aachen, Deutschland (Unknown); Psychotherapeutic outpatient clinic for children and adolescents, Catholic University Eichstätt-Ingolstadt, Germany (Unknown); Psychotherapeutic outpatient clinic for children and adolescents, University of Bamberg, Bamberg, Germany (Unknown); Center for Psychotherapie Bodensee (apb), Konstanz, Deutschland (Unknown); Child and Adolescent Outpatient Clinic (KJ-PAM), Universität Marburg, Marburg, Deutschland (Unknown); Child and Adolescent Psychiatric Services Thurgau, Switzerland (Unknown); Child and Adolescent Psychiatric Services St. Gallen, Switzerland (Unknown); Cantonal Hospital Winterthur, Switzerland (Unknown)
Responsible Party: Sponsor
Other Study IDs: BASEC 2025-01470
Record Dates: First submitted 2026-01-05; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: PTSD - Post Traumatic Stress Disorder; PTSD-Related Functional Impairment in Children and Adolescents
Keywords: PTSD; PTSS; Functional Impairment; PTSD-iMPACT; Validation; Posttraumatic stress disorder; Posttraumatic stress symptoms
MeSH Terms: conditions — Combat Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clinical population: The minimum sample size per Switzerland and Germany, respectively, will be n≥100 per cohort (n≥100 trauma-exposed children and adolescents aged 7-18, n≥100 caregivers of trauma-exposed children and adolescents aged 7-18; n≥100 caregivers of trauma-exposed children aged 3-6 years) to enable separate psychometric analyses for each country on a sufficient empirical basis. This corresponds, for each national sample (Switzerland and Germany), to a minimum of 100 trauma-exposed children and adolescents and a total of at least 200 caregivers. The maximum intended sample size is double these numbers. Consecutive data collection will continue at the participating study centers for 13 months (December 2025 - October 2026). As far as possible, every patient and/or caregiver who visits the participating clinical institutions or medical settings for the first time (inpatient or outpatient) will be invited to participate in the study.
- Non-clinical population: Only in Switzerland, a non-clinical sample will be recruited. The minimum sample size will be n≥100 trauma-exposed children and adolescents, and caregivers of trauma-exposed children and adolescents, per school type (Kindergarten [only caregivers], Primarschule [3rd grade or higher], Sekundarstufe [students and caregivers], Gymnasium [students until 18 and their caregivers], and Berufsschule [until 18 years]).
  Based on epidemiological data indicating that approximately 55% of Swiss adolescents report at least one potentially traumatic event, we plan to recruit a total minimum sample size of 200 children and adolescents and 200 caregivers in primary and secondary schools. An equally sized sample of 200 adolescents and 200 caregivers will be recruited in grammar schools (Gymnasium). In Berufsschulen, we aim to include 200 adolescents, while caregivers will not participate. For kindergartens, the recruitment target is 200 caregivers.

SUMMARY:
Population-based and clinical studies indicate that a substantial proportion of children and adolescents are exposed to one or more potentially traumatic events (PTEs) Approximately 16 % of those affected by childhood trauma go on to develop post-traumatic stress disorder (PTSD), with an even higher proportion experiencing subclinical levels of post-traumatic stress symptoms (PTSS). In Switzerland, over half of adolescents report exposure to at least one PTE, with 4.2 % meeting diagnostic criteria for PTSD. PTSD frequently impacts young people's social and educational functioning, often impairing their ability to engage in everyday life activities that are important or meaningful to them. Although the psychological consequences of PTSD are well documented, there is limited empirical understanding of how PTSS specifically affects day-to-day functioning in young people.

A key reason for this gap is the absence of a validated instrument specifically designed to assess PTSD-related functional impairment in children and adolescents. To address this need, the PTSD-iMPairment in Adolescent & Children's Capacity for Thriving (PTSD-iMPACT) measure was developed. This tool aims to systematically assess the extent of PTSD-related functional impairment in children and adolescents across key life domains, such as family, friends, school, apprenticeship, hobbies or media use.

The overall aim of this study is to evaluate the psychometric properties of the PTSD-iMPACT questionnaire in a clinical and in a non-clinical sample and to provide an internationally applicable standard instrument for the assessment of PTSD-related functional impairment in trauma-exposed children and adolescents.

In the long term, the aim is to ensure that the care and support provided to children and adolescents who experience difficulties in their daily lives due to post-traumatic stress symptoms are sustainably monitored and improved.

DETAILED DESCRIPTION:
The PTSD-iMPACT is designed to assess the severity of PTSD-related functional impairment across specific activities and tasks in multiple life domains.

The development of the PTSD-iMPACT followed a two-phase process. First, a systematic review was conducted to examine how existing PTSD-specific instruments, diagnostic interview modules, and general measures of functional impairment assess PTSD-related impairment in youth. The review revealed considerable heterogeneity in the domains assessed, frequent reliance on dichotomous response options, inconsistent scoring procedures, and a general lack of psychometric validation. Many instruments assessed functioning only at a global level, without capturing the specific nature or severity of difficulties within each domain. Furthermore, most relied on face validity and lacked demonstrated content validity, highlighting the need for a more methodologically sound tool.

In the second phase, qualitative interviews and focus groups were conducted (Cantonal Ethics Committee Zurich, Switzerland; BASEC-ID 2023-01290) with trauma-exposed children and adolescents (aged 7-18) who presented with at least moderate PTSS, as well as caregivers of children aged 1-18 with similar symptom profiles. Participants were recruited through clinical and social service settings. Data were analyzed using qualitative content analysis to identify relevant domains of functioning and specific challenges within those domains affected by PTSS. This conceptual framework informed item generation for the PTSD-iMPACT. Item refinement was carried out with input from clinical and research experts.

The final instrument includes both a self-report and caregiver-report version for children and adolescents aged 7-18, as well as a caregiver-version for children aged 3-6. It is designed to enhance clinical decision-making, improve diagnostic accuracy, and support outcome monitoring across diverse international contexts.

To ensure that the PTSD-iMPACT functions as a psychometrically sound and clinically meaningful assessment tool, validation across both clinical and non-clinical populations is essential and is therefore carried out in the present study. This process will allow for the evaluation of sensitivity, specificity, and broader applicability across varying levels of functional impairment, thereby supporting its use in both research and routine clinical practice.

The primary outcome will be the PTSD-iMPACT. The secondary outcomes for 7-18 year old children and adolescents include sociodemographic information, PTEs, PTSD, depression, anxiety, adjustment disorder, level of functioning, health-related quality of life, and regulation of emotional expression. The secondary outcomes for 3-6 year old children (caregiver-report) include sociodemographic information, PTEs, PTSD, depression, anxiety, oppositional behavior, adjustment disorder, stressor-related thoughts and worries, and health-related quality of life. Table 1 provides an overview of the constructs assessed and corresponding instruments used across participant groups.

Hypothesis and primary objective

The overall aim of this study is to evaluate the psychometric properties of the PTSD-iMPACT questionnaire in trauma-exposed children and adolescents. The specific aims of the present project are as follows:

1. To examine the reliability of the PTSD-iMPACT for children and adolescents aged 7 to 18 years. This includes the internal consistency of the self- and caregiver report, as well as the test-retest reliability of the PTSD-iMPACT, and the CATS-2 with a time span of two weeks.

   Hypothesis 1a: Internal consistency: We assume that the items of the PTSD-iMPACT self-report (7-18y) positively correlate with each other, as well as the items of the PTSD-iMPACT caregiver report (7-18y).

   Hypothesis 1b: Test-retest-reliability: We assume a positive correlation between the results of the first and second time of measurement of the PTSD-iMPACT (7-18y), as well as the CATS-2.
2. To examine the validity of the PTSD-iMPACT for children and adolescents aged 7 to 18 years, including the construct validity (convergent and divergent validity), the criterion validity (concurrent and predictive validity) and the factorial validity. Furthermore, we aim to determine an optimal cut-off value.

   Hypothesis 2a: Construct validity: We assume stronger positive correlations between the PTSD-iMPACT (7-18y) and the PTSD-specific instrument CATS-2 compared to its correlations with measures of general emotional and behavioral problems (IDQ, IAQ). Additionally, we expect the KIDSCREEN-10, which measures health-related quality of life, to show negative correlations with PTSD-iMPACT (7-18y). While not a direct measure of functional impairment, it captures aspects of well-being that are likely influenced by PTSD-related difficulties in daily life.

   Hypothesis 2b: Concurrent validity: We assume that the results of the PTSD-iMPACT (7-18y) positively correlate with the results of the Work and Social Adjustment Scale for Youth (WSAS-Y) and the universal 0-100 rating question "To what extent have the symptoms affected your child in daily life?".

   Hypothesis 2c: Predictive validity: We hypothesize that results of the PTSD-iMPACT (7-18y) differ between individuals with a normal, moderate, elevated and high PTSD symptomatology.

   Hypothesis 2d: Factorial validity: We assume that the theoretically and empirically derived structure of the PTSD-iMPACT (7-18y) is plausible (the factors reflect the subscales and the items of each subscale load onto their respective factors).
3. To examine the reliability of the PTSD-iMPACT for children aged 3 to 6 years. This includes the internal consistency of the caregiver report, as well as the test-retest reliability of the PTSD-iMPACT, and the CATS 3-6 with a time span of two weeks.

   Hypothesis 3a: Internal consistency: We assume that the items of the PTSD-iMPACT self-report (3-6y) positively correlate with each other, as well as the items of the PTSD-iMPACT caregiver report (3-6y).

   Hypothesis 3b: Test-retest-reliability: We assume a positive correlation between the results of the first and second time of measurement of the PTSD-iMPACT (3-6y), and the CATS 3-6
4. To examine the validity of the PTSD-iMPACT for children aged 3 to 6 years, including the construct validity (convergent and divergent validity), the criterion validity (concurrent and predictive validity) and the factorial validity. Furthermore, we aim to determine an optimal cut-off value.

   Hypothesis 4a: Construct validity: We assume stronger positive correlations between the PTSD-iMPACT (3-6y) and the PTSD-specific instrument CATS 3-6, compared to the correlations between results of the PTSD-iMPACT (3-6y) and questionnaires assessing general emotional and behavioral problems (CBCL subscales: anxiety, depression, oppositional behavior). Additionally, we expect the Pediatric Quality of Life Inventory (PedsQL) [22], which measures health-related quality of life, to show negative correlations with PTSD-iMPACT.

   Hypothesis 4b: Concurrent validity: We assume that the results of the PTSD-iMPACT negatively correlate with ad the universal 0-100 rating question "To what extent have the symptoms affected your child in daily life?".

   Hypothesis 4c: Predictive validity: We hypothesize, that results of the PTSD-iMPACT (3-6y) differ between individuals with a normal, moderate, elevated and high PTSD symptomatology.

   Hypothesis 4d: Factorial validity: We assume that the theoretically and empirically derived structure of the PTSD-iMPACT (3-6y) is plausible.

   Statistics and Methodology

   After the completion of data collection and prior to the statistical analysis of reliability and validity, a final integration of all measurement data from all participating centers will be conducted. Statistical analyses will be performed using R, SPSS and Mplus. All statistical analyses will be conducted using a two-sided significance level of α = 0.05. A minimum of 100 trauma-exposed participants per clinical cohort is deemed required.

   Statistical analysis for the PTSD-iMPACT (7-18 years) validation

   • Sample and items descriptives: Item description, item means, standard deviations, skewness, kurtosis, and range for both self- and caregiver report.

   Reliability
   * Internal consistency: Cronbach's alpha and McDonald's omega for PTSD-iMPACT (self- and caregiver report).
   * Test-retest reliability: The Intraclass Correlation Coefficient (ICC) will be calculated for PTSD-iMPACT, and the CATS-2.

   Validity

   Construct Validity:
   * Convergent validity: Correlations with the PTSD-specific instrument CATS-2, and the health-related quality of life measure (KIDSCREEN-10).
   * Divergent validity: Correlations with questionnaires assessing general emotional and behavioral problems (IDQ, and IAQ).

   Criterion Validity:
   * Concurrent validity: Correlations with the WSAS-Y. The universal 0-100 rating question will be used as an external criterion.
   * Predictive validity: Differentiation between individuals with a normal, moderate, elevated and high PTSD symptomatology (Mann-Whitney U test, Cohen's d). ROC analyses will be conducted to determine diagnostic accuracy (sensitivity, specificity). The optimal cut-off value will be determined using the Youden Index.

   Factorial Validity:

   • Confirmatory Factor Analysis (CFA): Examination of the theoretically and empirically derived structure of the questionnaire (subscales and item allocation). The CFA will assess whether the items load on the expected subscales, whether model fit indices are acceptable, and whether the correlations between factors are plausible.

   Statistical analysis for the PTSD-iMPACT (3-6 years) validation

   • Sample and items descriptives: Item description, item means, standard deviations, skewness, kurtosis, and range for caregiver-report.

   Reliability
   * Internal consistency: Cronbach's alpha and McDonald's omega for PTSD-iMPACT (caregiver report).
   * Test-retest reliability: The Intraclass Correlation Coefficient (ICC) will be calculated for PTSD-iMPACT, and the CATS 3-6.

   Validity

   Construct Validity:
   * Convergent validity: Correlations with the PTSD-specific instrument CATS 3-6and the health-related quality of life measure (PedsQL).
   * Divergent validity: Correlations with questionnaires assessing general emotional and behavioral problems (CBCL subscales: anxiety, depression, oppositional behavior).

   Criterion Validity:
   * Concurrent validity: Correlations with the PedsQL. The universal 0-100 rating question will be used as an external criterion.
   * Predictive validity: Differentiation between individuals with a normal, moderate, elevated and high PTSD symptomatology (Mann-Whitney U test, Cohen's d). ROC analyses will be conducted to determine diagnostic accuracy (sensitivity, specificity). The optimal cut-off value will be determined using the Youden Index.

   Factorial Validity:

   • Confirmatory Factor Analysis (CFA): Examination of the theoretically and empirically derived structure of the questionnaire (subscales and item allocation). The CFA will assess whether the items load on the expected subscales, whether model fit indices are acceptable, and whether the correlations between factors are plausible.

   Handling of missing data

   Missing data will be addressed using the Multiple Imputation (MI) method in R, which generates multiple plausible datasets by imputing missing values based on observed data. This approach allows for the inclusion of all available data without case-wise deletion, under the assumption that data are missing completely at random (MCAR) or missing at random (MAR). The analyses will be conducted across all imputed datasets, and the results will be pooled to account for the variability introduced by imputation.

   To assess the potential impact of missing follow-up data, a sensitivity analysis will be performed by comparing results from the pooled imputed datasets with a complete-case analysis, including only participants who completed both measurement points. If substantial differences between these approaches emerge, this may suggest systematic dropout (i.e., data missing not at random [MNAR]), which will be considered in the interpretation of the findings.

   Study Design

   This study employs a quantitative and confirmatory study design. The confirmatory nature of the study reflects its primary objective - to test predefined hypotheses regarding the psychometric properties of the PTSD-iMPACT measure. Furthermore, the planned project is designed as an international multicenter validation study of the PTSD-iMPACT measure with study sites in Switzerland and Germany. Depending on the individual study site and its available resources, the design is either cross-sectional or longitudinal. The coordinating study center is the Department of Psychosomatics and Psychiatry at the University Children's Hospital Zurich, Switzerland. The coordinating center is responsible for data management and statistical analysis. Recruitment and data collection will be conducted in a clinical and non-clinical sample to increase the generalizability of the findings. The inclusion of both clinical and non-clinical samples is strategically designed to validate the PTSD-iMPACT across a wide range of PTSS severity, functional impairments, and sociodemographic characteristics, thereby strengthening the external validity of the instrument.

   The Project is structured in three phases:

   Phase 1

   Based on results of a systematic review, qualitative interviews/ focus groups, and expert rating, as well as clinical experience in treating traumatized children and adolescents, an English-language reference version of the PTSD-iMPACT measure was developed.

   The PTSD-iMPACT measure is available in the following three versions
   * Self-report by children and adolescents aged between 7 and 18
   * Caregiver-report of children and adolescents aged between 7 and 18
   * Caregiver-report of children and adolescents aged between 3 and 6

   In a first step, two independent forward translations into the respective language (German), a consensus procedure in case of deviations, an independent backward translation into the source language (American English) will be conducted. If necessary, a final round for a consensus procedure in case of deviations from the original version will be created and carried out.

   Phase 2

   The aim of this phase is to collect data and test the psychometric properties in different clinical settings in both Switzerland and Germany and in a non-clinical setting (schools) in Switzerland.

   Clinical population:

   Once the minimum number of cases for psychometric analyses has been reached (n≥100 per country and cohort), the data will be analyzed at the coordinating study center to determine the psychometric quality of the new measurement instrument in clinical populations between the ages of 7 and 18 (self- and caregiver-report) and between the ages of 3 and 6 (caregiver-report). In total, each participant (children/adolescents and caregiver) will complete the whole questionnaire battery once and two weeks later a second questionnaire battery, including only PTSD (CATS-2/ CATS 3-6, PTSD-related functional impairment (PTSD-iMPACT), and adjustment disorder (IADQ-CA/IADQ-CA 3-6). If desired, participants may choose to take part in only the first assessment. The effort required is approx. 40 minutes for the first assessment and approx. 15 minutes for the second assessment.

   Non-clinical setting (Switzerland only):

   Once the minimum number of cases for psychometric analyses has been reached (n≥100 trauma-exposed children and adolescents, or caregivers of trauma-exposed children and adolescents per type of school (Kindergarten [only caregivers], Primarschule [3rd grade or higher], Sekundarstufe [students and caregivers), Gymnasium (students until 18 and their caregivers, and Berufsschule [until 18 years]), the data will be analyzed at the coordinating study center to determine the psychometric quality of the new measurement instrument in non-clinical populations between the ages of 7 and 18 (self- and caregiver-report) and between the ages of 3 and 6 (caregiver-report). In total, each participant (children/adolescents and caregivers) will complete the questionnaire battery once. The effort required is approx. 40 minutes. Questionnaire data will be collected using an online secured survey tool, namely REDCap [20], hosted by the University Children's Hospital Zurich. Participants will enter all information directly into REDCap or, if schools are unable to provide computers or tablets, via paper-and-pencil questionnaires.

   Phase 3

   Once the data analysis has been completed, the final PTSD-iMPACT measure will be disseminated as a free download in paper-and-pencil format. In addition, a short, easy-to-understand manual with examples of use and evaluation will be developed. The manual will be made available to promote the use of the questionnaire in routine care (outpatient and inpatient).

   Expected Biases

   Language distortion: The majority of participants in this study will primarily consist of children, adolescents, and caregivers with a sufficient understanding of the German language. Therefore, the sample will predominantly be comprised of individuals who are fluent in German. Consequently, the overall population of exposed children and adolescents might not be fully represented in the present study. The aforementioned bias will be taken into account when the results are interpreted.

   Self-selection: There could potentially be a risk that trauma-exposed children and adolescents and caregivers of trauma-exposed children and adolescents who have higher functioning levels both mentally and physically, are more inclined to participate and thus, certain domains of functional impairment and corresponding difficulties will be rated as more or less important. This bias will be considered when discussing the results. Further, a potential bias in the planned study is the distinction between individuals with and without PTEs, which could influence data interpretation. To mitigate this, this classification will only be made after the data collection.

   Recruitment process

   Different recruitment procedures will be implemented and conducted for different study sites.

   Switzerland - clinical institutions

   As far as possible, every patient and/or caregiver who visits the participating Swiss clinical institutions or medical settings for the first time (inpatient or outpatient) will be invited to participate in the study. The treating mental health specialist will inform the patients and their caregivers verbally about the study. In case of interest, the treating mental health specialist obtains verbal consent to forward their contact information (Name, Surname, phone number, e-mail address) to the study coordinator and give out study information (including consent form). The coordinating research team contacts the potentially participants and provides detailed information about the study (i.e., purpose, duration, timeline, voluntary nature, potential risks, benefits). Signed consent forms are returned electronically by email. After reception, adolescents between 12 and 18 years and caregivers of children/adolescents between 3 and 18 years receive a personalized but de-identified REDCap link via email to complete the initial questionnaire battery. A follow-up link will be sent two weeks later to assess test-retest reliability. For children between 7 and 11 years, the coordinating research team will schedule a phone or video call via Microsoft Teams to assist with completing the initial questionnaire battery, followed by a second call two weeks later to support completion of the follow-up battery. This approach ensures standardization of administration while providing age-appropriate guidance. Patients /caregivers in the study can choose whether their findings is supposed to be reported to their treating mental health specialist. If desired a standardized brief report, entailing the overarching results of the questionnaires, will be send by the study coordinator to the local study leader, respectively, which then distributes the report to the treating mental health specialist at site.

   Recruitment by the Child Protection Group of the University Children's Hospital Zurich follows the same procedure as described for psychotherapeutic settings, with two exceptions: recruitment is conducted not by a psychotherapist, but by the designated person in charge of the Child Protection Group, and there is no option for questionnaire results to be shared with a treating psychotherapist, as these participants are not recruited within a psychotherapeutic context.

   Switzerland - medical settings

   At the University Children's Hospital, medical patients and their caregivers, who were referred to the emergency department and who have signed the hospital's general research consent form will be recruited. Recruitment takes place approximately four weeks after referral. They will be contacted via telephone by trained study personnel of the research team, who provide detailed information about the study (i.e., purpose, duration, timeline, voluntary nature, potential risks, benefits). If they are interested in participating afterwards, they receive study information and informed consent. Signed consent forms are returned electronically by email. After reception, adolescents between 12 and 18 years and caregivers of children/adolescents between 3 and 18 years receive a personalized but de-identified REDCap link to complete the initial questionnaire battery. A follow-up link will be sent two weeks later to assess test-retest reliability. For children between 7 and 11 years, the coordinating research team will schedule a phone or video call via Microsoft Teams to assist with completing the initial questionnaire battery, followed by a second call two weeks later to support completion of the follow-up battery. This approach ensures standardization of administration while providing age-appropriate guidance.

   Switzerland - Students/ caregiver of kindergartners and students (non-clinical population)

   Data of students (all German-speaking cantons) and caregivers of kindergartners (all German-speaking cantons) and students (all German-speaking cantons) will be collected. No second assessment two weeks later will take place in the non-clinical population.

   The survey introduction explicitly states that individuals should not participate if they have already taken part in the study through clinical recruitment, lack sufficient German language skills, or fall outside the eligible age range. The same questionnaires and socio-demographic measures used in the clinical sample will be applied. Participation takes approximately 40 minutes. No follow-up assessment is planned for the non-clinical sample.

   Kindergartens

   All kindergartens in the German-speaking part of Switzerland will be invited to participate in the planned study. In case of participation, a REDCap link to the anonymous questionnaires will be send to the caregivers by the teachers via email list, respectively. The start of the survey provides information about the study (purpose, content, handling of data). At the end of the introduction, caregivers have to mark actively if they would like to participate (or not). In case of participation, they subsequently fill out the questionnaire. In case of no participation, the survey ends.

   Schools

   Schools in German-speaking cantons will be invited to participate in the planned study. Data collection on site will be coordinated in advance with school leadership and teachers. Whenever possible, data collection will be conducted in the classroom setting, as this provides an optimal environment for participant safety and support. Children and adolescents grade 3 or above will complete the questionnaire battery during class hours. Two weeks before data collection, students/caregivers will receive an information letter about the study. The letter outlines the study's purpose and content and provides advance notice of the upcoming assessment. Further, the letter entails a brief consent form, allowing children and their caregivers to indicate whether the child would like/ is allowed to participate. Adolescents aged 14 and older may sign the form themselves. Completed forms will be returned to the teacher. On the day of data collection, the teacher will verify which students have consented to participate-without disclosing any names to the research team. Students who do not participate, or who have already taken part in the clinical arm of the study, will be given alternative activities during the survey period. On assessment day, three or more trained members of the research team will be present during the assessment, supervising small groups to ensure comprehension and provide assistance if needed. Also, the research team will keep a watching eye on the students to detect any signs of stress or discomfort early on. Participants will complete the questionnaire either digitally (on school-provided tablets or computers) or using a paper-and-pencil format. Members of the research team will each have a copy of the questionnaires. In case of questions, students student can point out the item to the research team, which then uses their copy as a basis to answer the questions. This ensures complete anonymity and confidentiality. Following completion of the questionnaire, the students received an information sheet with a list of easily accessible institutions that provided help for mental health problems. At the start of the session, students will be clearly instructed not to write their names on the questionnaires. In case of a student reaching out to the research team after assessment (e.g., because of emotional distress), no link can be made to their survey data. The study team will not inquire about answers to specific questions. This approach allows for an individualized follow-up without compromising anonymity or data protection. Students will be informed that participation is completely voluntarily and that they can end the assessment at any point (e.g., in case of emotional distress). In case of severe emotional distress, students will be made aware of easily accessible institutions that provided help for mental health problems in children and adolescents.

   Caregivers of children and adolescent will receive a REDCap link to the questionnaire battery from the teacher by email, and if interested, complete the survey at home. If classroom-based data collection is not feasible for adolescents (aged 12-18), they will be provided with a REDCap survey link to complete the questionnaire independently outside of school hours. The link will be sent by the teacher. All participants will receive contact information for the emergency psychiatric services (KANT) at the Psychiatric University Hospital Zurich, which are available 24/7 in cases of acute psychological distress. Additionally, contact details for the study team will be provided for participants who experience elevated distress and wish to seek support.

   Germany - clinical institutions or medical settings

   The German local study site University Clinic for Child and Adolescent Psychiatry, Psychosomatics, and Psychotherapy, Carl von Ossietzky University of Oldenburg, Germany acts subordinate further as co-coordinating center for the following German clinical study sites under Dr. M. Vasileva.

   Following approval of the Swiss application by the Cantonal Ethics Committee Zurich, the German co-coordinating study site will submit the approval to its respective local ethics committee. Depending on local resources and funding available, the following recruitment/ data collection strategies will be applied at the German study sites:

   Recruitment Strategy A As far as possible, every patient and/or caregiver who visits the participating clinical institutions or medical settings for the first time (inpatient or outpatient) will be invited to participate in the study. The treating mental health specialist will inform the patients and their caregivers verbally about the study. In case of interest, the treating mental health specialist obtains written consent (equivalent to an Authorization for Release of Psychotherapy Information) that allows the mental health specialist to forward their contact information (Name, Surname, phone number, e-mail address) to the study coordinator M.Sc. A. Vogt via HIN-mail and give out study information (including consent form). The document will be filed in the patient record. The coordinating research contacts the potentially participants and provides detailed information about the study (i.e., purpose, duration, timeline, voluntary nature, potential risks, benefits). Signed consent forms are returned electronically by email. After reception, adolescents between 12 and 18 years and caregivers of children/adolescents between 3 and 18 years receive a personalized but de-identified REDCap link to complete the initial questionnaire battery. A follow-up link will be sent two weeks later to assess test-retest reliability. For children between 7 and 11 years, the coordinating research team will schedule a phone or video call via Microsoft Teams to assist with completing the initial questionnaire battery, followed by a second call two weeks later to support completion of the follow-up battery. This approach ensures standardization of administration while providing age-appropriate guidance. Patients/ caregivers in the study can choose whether their findings is supposed to be reported to their treating mental health specialist. If desired a standardized brief report, entailing the overarching results of the questionnaires, will be send by the Swiss study coordinator A. Vogt to the local study leader, respectively, which then distributes the report to the treating mental health specialist at site.

   Recruitment Strategy B As far as possible, every patient and/or caregiver who visits the participating clinical institutions or medical settings for the first time (inpatient or outpatient) will be invited to participate in the study. The treating mental health specialist will inform the patients and their caregivers verbally about the study and hand out a flyer about the study, including a generalized link to the questionnaire battery on REDCap. Interested caregivers (of children of all age groups) and adolescents aged 12-18 years will access and complete the questionnaire independently. Children aged 7 to 11 years will not be included in this recruitment strategy. Since the link is general, anonymity is guaranteed. Data can therefore not be shared with the treating psychotherapeutic professional. The respective version of the study information is shown at the start of the questionnaire and participants have to sign the consent form in digital form. Participants will not complete a follow-up questionnaire battery.

   Recruitment Strategy C As far as possible, every patient and/or caregiver who visits the participating clinical institutions or medical settings for the first time (inpatient or outpatient) will be invited to participate in the study trough the local study site leaders and their research team. Informed consent will be obtained and data will be collected through the Swiss REDCap server and tool from the University-Children's Hospital Zurich via tablet at the German study site. Data collection will be anonymously. Informed consent will be collected through the local study site leader or a member of their research team electronically via REDCap before administering the questionnaires.

   No procedure relating to the project will be carried out before consent has been given by the participant. Only data collected after consent is given will be used for analysis. Any contact details shared with the study team will be deleted if the potential participants decide not to take part in the study.

ELIGIBILITY:
Clinical population

Inclusion Criteria:

* Use of (mental) health services at a participating study center.
* Children and adolescents between 7 and 18 years / caregivers of children and adolescents between 3 and 18 years
* Sufficient knowledge of the German language
* Signed consent form (7-18 years: patient and caregiver; 3-6 years: caregivers)

Exclusion Criteria:

* Children and adolescents under 7 or over 18 years / caregivers of children and adolescents under 3 or over 18 years
* Not sufficient knowledge of the German language
* No signed consent form (7-18 years: patient and/or caregiver; 3-6 years: caregivers)

Non-clinical population Only recruited in Switzerland.

Inclusion Criteria:

* Students between 3rd grade and 18 years / caregivers of kindergarteners and students up until 18 years
* Sufficient knowledge of the German language

Exclusion Criteria:

* Students 2nd grade or lower and over 18 years / caregivers of children not yet in Kindergarten and students over 18 years
* No sufficient knowledge of the German language

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Clinical sample:
  As far as possible, every patient and/or caregiver who visits the participating clinical institutions or medical settings in Switzerland and Germany for the first time (inpatient or outpatient) will be invited to participate in the study.
  Non-clinical sample:
  Data of students (all German-speaking cantons) and caregivers of kindergartners (all German-speaking cantons) and students (all German-speaking cantons) will be collected.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
PTSD-iMPACT (newly developed questionnaire) | Baseline and Follow-up two weeks later. In nonclinical samples, data will be only assessed at Baseline.
  Children and Adolescents aged 7 to 18 years:
  Self-report and caregiver-report.
  The following domains are assessed:
  * Family - Living together (5 items)
  * Family - Contact without living together (4 items)
  * Friends/Peers (5 items)
  * School (5 items)
  * Work/Vocational Program/Apprenticeship (5 items)
  * Hobbies/Fun (3 items)
  * Dating/Romantic Relationships (3 items)
  * Getting around and joining in (2 items)
  * Health/Self-Care (5 items)
  * Media Use (1 item)
  Children aged 3 to 6 years:
  Caregiver-report.
  The following domains are assessed:
  * Family - Living together (5 items)
  * Family - Contact without living together (4 items)
  * Friends/Peers (4 items)
  * Daycare/Preeschool/Kindergarten/School (3 items)
  * Playing/Fun (2 items)
  * Public places (1 item)
  * Health/Self-Care (2 items)
  * Media Use (1 item)

SECONDARY OUTCOMES:
Potentially traumatic events (PTE) (Children and adolescents aged 7 to 18 years) | Baseline and Follow-up two weeks later. In nonclinical samples, data will be only assessed at Baseline.
  Child and Adolescent Trauma Screen (CATS 2)
PTSD (Children and adolescents aged 7 to 18 years) | Baseline and Follow-up two weeks later. In nonclinical samples, data will be only assessed at Baseline.
  Child and Adolescent Trauma Screen (CATS 2)
Depression (Children and adolescents aged 7 to 18 years) | Baseline
  International Depression Questionnaire (IDQ)
Anxiety (Children and adolescents aged 7 to 18 years) | Baseline
  International Anxiety Questionnaire (IAQ
Quality of life (Children and adolescents aged 7 to 18 years) | Baseline
  KIDSCREEN-10
Functioning (Children and adolescents aged 7 to 18 years) | Baseline
  Work and Social Adjustment Scale-Youth (WSAS-Y)
Adjustment disorder (both children 3-6 and 7-18years) | Baseline and Follow-up two weeks later. In nonclinical samples, data will be only assessed at Baseline.
  International Adjustment Disorder Questionnaire - Child and Adolescent (IADQ-CA)
Regulation of Emotional Expression (Children and adolescents aged 7 to 18 years) | Baseline
  Flexible Regulation of Emotional Expression Scale (FREE)
Potentially traumatic events (Children aged 3 to 6 years) | Baseline and Follow-up two weeks later. In nonclinical samples, data will be only assessed at Baseline.
  Child and Adolescent Trauma Screen (CATS 3-6)
PTSD (Children aged 3 to 6 years) | Baseline and Follow-up two weeks later. In nonclinical samples, data will be only assessed at Baseline.
  Child and Adolescent Trauma Screen (CATS 3-6)
Behavioral Problems (Children aged 3 to 6 years) | Baseline
  Child Behavior Checklist (CBCL 1½-5; DSM-5 subscales: affective problems, anxiety problems, oppositional defiant problems)
Quality of Life (Children aged 3 to 6 years) | Baseline
  Pediatric Quality of Life Inventory (PedsQL)
Stressor-related Thoughts and Worries (Children aged 3 to 6 years) | Baseline
  Preschooler Stressor-related Thoughts and Worries scale (PSTWS)
PTSD (Caregiver of children aged 3 to 6) | Baseline and Follow-up two weeks later. In nonclinical samples, data will be only assessed at Baseline.
  International Trauma Questionnaire (ITQ)
Trauma Exposure (Caregiver of children aged 3 to 6) | Baseline and Follow-up two weeks later. In nonclinical samples, data will be only assessed at Baseline.
  International Trauma Exposure Measure (ITEM)

OTHER OUTCOMES:
Sociodemographic information of Children and adolescents | Baseline
  Age (in years), gender/sex, type of school, school grade, number of siblings, country of origin of child, country of origin of caregiver, employment of caregiver, living situation, satisfaction with academic performance, psychotherapy
Sociodemographic information of caregivers | Baseline
  Age (in years) of child and caregiver, gender/sex child and caregiver, type of school child, school grade child, number of siblings child, country of origin of caregiver, education of caregiver, employment of caregiver, child's living situation, child's satisfaction with academic performance, psychotherapy child

CONTACTS AND LOCATIONS:
Locations (11):
- Germany (7):
  - Traumaambulanz, Universitätsklinikum Aachen, Aachen
  - Otto-Friedrich-Universität Bamberg, Bamberg
  - Lehrstuhl für Klinische Psychologie und Kinder- und Jugendlichenpsychotherapie, Katholische Universität Eichstätt-Ingolstadt, Eichstätt
  - Zentrum für Psychotherapie Bodensee (apb), Konstanz
  - Kinder- und Jugendlichen-Psychotherapie-Ambulanz (KJ-PAM) Marburg, Marburg
  - Universitätsklinik für Kinder- und Jugendpsychiatrie, Psychosomatik und Psychotherapie Carl von Ossietzky Universität Oldenburg, Oldenburg
  - Child and Adolescent Psychiatry Ulm University, Ulm
- Switzerland (4):
  - Child and Adolescent Psychiatric Services Thurgau, Frauenfeld
  - • Parent-Child Consultation 0-5 of The Child and Adolescent Psychiatric Services St. Gallen, Sankt Gallen
  - Cantonal Hospital Winterthur, Winterthur
  - University Children's Hospital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hyland P, Karatzias T, Shevlin M, McElroy E, Ben-Ezra M, Cloitre M, Brewin CR. Does requiring trauma exposure affect rates of ICD-11 PTSD and complex PTSD? Implications for DSM-5. Psychol Trauma. 2021 Feb;13(2):133-141. doi: 10.1037/tra0000908. Epub 2020 Sep 10. PMID 32915045
- [Background] Cloitre M, Shevlin M, Brewin CR, Bisson JI, Roberts NP, Maercker A, Karatzias T, Hyland P. The International Trauma Questionnaire: development of a self-report measure of ICD-11 PTSD and complex PTSD. Acta Psychiatr Scand. 2018 Dec;138(6):536-546. doi: 10.1111/acps.12956. Epub 2018 Sep 3. PMID 30178492
- [Background] Haag AC, Cha CB, Noll JG, Gee DG, Shenk CE, Schreier HMC, Heim CM, Shalev I, Rose EJ, Jorgensen A, Bonanno GA. The Flexible Regulation of Emotional Expression Scale for Youth (FREE-Y): Adaptation and Validation Across a Varied Sample of Children and Adolescents. Assessment. 2023 Jun;30(4):1265-1284. doi: 10.1177/10731911221090465. Epub 2022 May 5. PMID 35510578
- [Background] Vasileva, M., Marsac, M. L., Alisic, E., Cobham, V. E., Davis, S. H., Donovan, C., ... & De Young, A. (2022). Preschooler stressor-related thoughts and worries during the COVID-19 pandemic: Development and validation of a caregiver-report instrument. Traumatology.
- [Background] Vogt, A., Berliner, L., Sachser, C., Theimer, K., Landolt, M. A., & Bartels, L. (2025). PTSD-iMPairment in Adolescent & Children's capacity for Thriving (PTSD-iMPACT). [Unpublished measurement instrument]. University Children's Hospital Zurich.
- [Background] Varni JW, Seid M, Kurtin PS. PedsQL 4.0: reliability and validity of the Pediatric Quality of Life Inventory version 4.0 generic core scales in healthy and patient populations. Med Care. 2001 Aug;39(8):800-12. doi: 10.1097/00005650-200108000-00006. PMID 11468499
- [Background] Kristensen S, Henriksen TB, Bilenberg N. The Child Behavior Checklist for Ages 1.5-5 (CBCL/1(1/2)-5): assessment and analysis of parent- and caregiver-reported problems in a population-based sample of Danish preschool children. Nord J Psychiatry. 2010 May 4;64(3):203-9. doi: 10.3109/08039480903456595. PMID 20085433
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Jassi A, Lenhard F, Krebs G, Gumpert M, Jolstedt M, Andren P, Nord M, Aspvall K, Wahlund T, Volz C, Mataix-Cols D. The Work and Social Adjustment Scale, Youth and Parent Versions: Psychometric Evaluation of a Brief Measure of Functional Impairment in Young People. Child Psychiatry Hum Dev. 2020 Jun;51(3):453-460. doi: 10.1007/s10578-020-00956-z. PMID 32006302
- [Background] Ravens-Sieberer U, Herdman M, Devine J, Otto C, Bullinger M, Rose M, Klasen F. The European KIDSCREEN approach to measure quality of life and well-being in children: development, current application, and future advances. Qual Life Res. 2014 Apr;23(3):791-803. doi: 10.1007/s11136-013-0428-3. Epub 2013 May 18. PMID 23686556
- [Background] Redican E, Sachser C, Berliner L, Pfeiffer E, Martsenkovskyi D, Hyland P, Ben-Ezra M, Shevlin M. Development and validation of the caregiver-report version of the international depression questionnaire (IDQ-CG) and international anxiety questionnaire (IAQ-CG). Eur Child Adolesc Psychiatry. 2025 Jan;34(1):297-305. doi: 10.1007/s00787-024-02495-7. Epub 2024 Jun 18. PMID 38888671
- [Background] Bartels, L., Berliner, L., Landolt, M., Shevlin, M., & Sachser, C. (2025). International Adjustment Disorder Questionnaire - Child and Adolescent Version (IADQ-CA) [Unpublished questionnaire]. University Children's Hospital Zurich.
- [Background] Sachser C, Berliner L, Holt T, Jensen TK, Jungbluth N, Risch E, Rosner R, Goldbeck L. International development and psychometric properties of the Child and Adolescent Trauma Screen (CATS). J Affect Disord. 2017 Mar 1;210:189-195. doi: 10.1016/j.jad.2016.12.040. Epub 2016 Dec 27. PMID 28049104
- [Background] Nilsson D, Davelid I, Ledin S, Svedin CG. Psychometric properties of the Child and Adolescent Trauma Screen (CATS) in a sample of Swedish children. Nord J Psychiatry. 2021 May;75(4):247-256. doi: 10.1080/08039488.2020.1840628. Epub 2020 Nov 8. PMID 33164607
- [Background] Sachser C, Berliner L, Risch E, Rosner R, Birkeland MS, Eilers R, Hafstad GS, Pfeiffer E, Plener PL, Jensen TK. The child and Adolescent Trauma Screen 2 (CATS-2) - validation of an instrument to measure DSM-5 and ICD-11 PTSD and complex PTSD in children and adolescents. Eur J Psychotraumatol. 2022 Aug 1;13(2):2105580. doi: 10.1080/20008066.2022.2105580. eCollection 2022. PMID 35928521
- [Background] Vogt, A. J., Landolt, M. A., Skjærvø, I., Hermann, R. M.m Pfeiffer, E., Sachser, C., & Bartels, L. (in preparation) Assessment of Posttraumatic Stress-Related Functional Impairment in Children and Adolescents: a Systematic Review.
- [Background] Landolt MA, Schnyder U, Maier T, Schoenbucher V, Mohler-Kuo M. Trauma exposure and posttraumatic stress disorder in adolescents: a national survey in Switzerland. J Trauma Stress. 2013 Apr;26(2):209-16. doi: 10.1002/jts.21794. Epub 2013 Mar 13. PMID 23494743